CLINICAL TRIAL: NCT02940899
Title: Fit Families Program for Children With Autism
Brief Title: Syracuse University Fit Families Program: Autism
Acronym: SUFFP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Collaborators: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Luis Columna, Associate Professor, Syracuse University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 28491
Record Dates: First submitted 2016-06-03; First posted 2016-10-21 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Syracuse University Fir Families Program (SUFFP) (Active Comparator): SUFFP is a randomized control trial comparing two groups of families of children with autism spectrum disorders. 20 families participated in the intervention program
  Interventions: Other: Intervention: Syracuse University Fir Families Program (SUFFP)
- Control: Syracuse University Fir Families Program (SUFFP) (Active Comparator): 20 families served as a wait-list control group. The control group will fill out the same pre and post measures as the intervention families (membership in the control vs. intervention group will be selected semi-randomly such that the average age of each of the two groups is equal), which will allow us to tease apart the effects of development vs. those related to the intervention.
  Interventions: Other: Intervention: Syracuse University Fir Families Program (SUFFP)

INTERVENTIONS:
Other: Intervention: Syracuse University Fir Families Program (SUFFP) — The SUFFP (Syracuse University Fit Families Program) is a randomized clinical trial, were 40 children with autism spectrum disorders ages 5-11 and at least one parent were randomly assigned to one of two group-based conditions; interventions or a control wait list group.

SUMMARY:
Syracuse University Fit Families is designed to increase the activity level and frequency of the children through modified activities using adapted equipment and, importantly, to increase the families' comfort level in having their children participate in a variety of physical activities, including team and individual sports.

DETAILED DESCRIPTION:
Syracuse University Fit Families is designed to increase the activity level and frequency of the children through modified activities using adapted equipment and, importantly, to increase the families' comfort level in having the children participate in a variety of physical activities, including team and individual sports. By increasing physical activity levels, investigators can reduce sedentary behaviors that lead to conditions such as obesity and cardiovascular diseases. The investigators will provide a series of workshops that will also teach children and families how to access nearby facilities and modify familiar activities, resulting in health benefits for all. Children, and parents will be involved in developmentally designed, land-based and aquatic physical activities. Parents will be engage in vibrant discussions with professionals and other parents who share similar experiences.

Services provided through the Syracuse University Fit families program are designed to improve the emotional, social and physical well-being of the participants. This program will include 1) educational seminars for parents on topics that improve awareness, advocacy, and access to community services; 2) inclusive games and modified sports for children, and parents to improve self-awareness, social interactions, and physical fitness; 3) individual consultation with physical activity professionals to address children's and families' social and recreational needs; and 4) opportunities for social networking for families participating in the program, including mentoring of youth by adapted sports athletes.

The project is proposed to run from November 2015 through June 2017. Five one-day workshops will be offered annually to participants covering topics of: 1) sensory integration, 2) communication, 3) motor development and physical activity; 4) aquatic; and 5) sport opportunities (individual and team sport). As part of program evaluation, the investigators will be conducting measurements on parents (e.g., quality of life, physical activity levels) and children (e.g., social communication, sensory behaviors, quality of life, physical activity levels, blood pressure). The investigators will assess these in a pre-post fashion in order to determine whether the program has led to generalized improvements in these areas. The testing procedure requires minimal invasion and it is not overwhelming for the participants. The investigators have implemented similar procedures in previous programs.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of autism spectrum disorders
* Children with autism spectrum disorders 5-11 years old
* Must be ambulatory
* Must be able to follow verbal or picture directions with support.
* Must not exhibit aggressive behavior.

Exclusion Criteria:

* Children with autism spectrum disorders younger than 4-11 years old
* Children with autism spectrum disorders older than 11 years old

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Physical Activity | Two years
  To assess physical activity levels among families of children with autism spectrum disorders. This outcome will be measured by counting steps by day using accelerometry.

SECONDARY OUTCOMES:
Motor skills of Parents and Children | Two years
  To asses the motor skills of parents and children with autism spectrum disorders. This outcome will be measured using the Test of Gross Motor Development 2.
Adaptive behavior | Two years
  To asses adaptive behavior of children with autism spectrum disorders. This outcome will be measured using the Vinland Adaptive Behavior Scales.
Reported Behavior Problems | Two years
  To asses is there a change in parents' reported behavioral problems of children with autism spectrum disorders as a result of the intervention. This outcome will be measured using the Behavior Assessment System for Children (BASC 2).
Sensory Processing | Two years
  To asses is there a change in in sensory processing as a result of the intervention. This outcome will be measured using the Sensory Profile (Dunn 1999).
Quality of Life of Parents of Children with Autism Spectrum Disorders | Two years
  To asses the quality of life children with autism spectrum disorders. This outcome will be measured using self reports.
Physical Activity Experiences | Two years
  To asses parents' experiences regarding physical activity. This will be measured using qualitative parent interviews.
Physical Activity Experiences | Two years
  To asses parents' experiences regarding physical activity. This will be measured using quantitative parent reports.
Cardiovascular Health | Two years
  Examine the effect of Fit Families on arterial stiffness in children with ASD. This will be derived from brachial pressure waveforms obtained via an oscillometric cuff.
Cardiovascular Health | Two years
  Examine the effect of Fit Families on central blood pressure in children with ASD. This will be derived from brachial pressure waveforms obtained via an oscillometric cuff.
Cardiovascular Health | Two years
  Examine the effect of Fit Families on arterial stiffness in the parents of children with ASD. This will be derived from brachial pressure waveforms obtained via an oscillometric cuff.
Cardiovascular Health | Two years
  Examine the effect of Fit Families on central blood pressure in the parents of children with ASD. This will be derived from brachial pressure waveforms obtained via an oscillometric cuff.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Columna, Ph.D, Principal Investigator — Syracuse University
Locations (1):
- Syracuse University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No